CLINICAL TRIAL: NCT06742424
Title: Efficacy and Safety of PD-L1 Antibody Combined With Bevacizumab and Hepatic Arterial Infusion Chemotherapy in Advanced Unresectable Hepatocellular Carcinoma With Extrahepatic Metastases: A Single-Arm, Prospective, Phase II Clinical Study
Brief Title: PD-L1 Antibody + Bevacizumab With Hepatic Arterial Infusion Chemotherapy for Advanced HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Wentao Wang, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024(2134)
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Hepato Cellular Carcinoma (HCC)
Keywords: HAIC; PD-L1; Bevacizumab; extrahepatic metastases
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-L1 Antibody + Bevacizumab + HAIC-FOLFOX (Experimental): Participants will receive:
  * PD-L1 antibody 1200mg intravenously every 3 weeks
  * Bevacizumab 15mg/kg intravenously every 3 weeks
  * HAIC-FOLFOX regimen (up to 6 cycles) consisting of:
    * Oxaliplatin 130 mg/m² via hepatic arterial infusion over 3 hours
    * Leucovorin 400 mg/m² via hepatic arterial infusion over 2 hours
    * Fluorouracil 400 mg/m² bolus via hepatic arterial infusion at hour 5, followed by 2400 mg/m² continuous hepatic arterial infusion over 46 hours
    * HAIC treatment repeats every 3 weeks for up to 6 cycles After completion of HAIC, participants will continue to receive PD-L1 antibody and bevacizumab until disease progression, unacceptable toxicity, or up to 24 months of treatment. Tumor assessments will be performed every 9 weeks for the first 48 weeks, then every 12 weeks thereafter.
  Interventions: Drug: PD-L1 antibody; Drug: Bevacizumab; Procedure: HAIC-FOLFOX

INTERVENTIONS:
Drug: PD-L1 antibody — 1200mg intravenously every 3 weeks
Drug: Bevacizumab — 15mg/kg intravenously every 3 weeks
Procedure: HAIC-FOLFOX — Oxaliplatin 130 mg/m² via hepatic arterial infusion over 3 hours Leucovorin 400 mg/m² via hepatic arterial infusion over 2 hours Fluorouracil 400 mg/m² bolus via hepatic arterial infusion at hour 5, followed by 2400 mg/m² continuous hepatic arterial infusion over 46 hours HAIC treatment repeats every 3 weeks for up to 6 cycles

SUMMARY:
This is a single-arm, phase II clinical trial evaluating the safety and efficacy of PD-L1 antibody combined with bevacizumab and hepatic arterial infusion chemotherapy (HAIC) for patients with advanced unresectable hepatocellular carcinoma (HCC) with extrahepatic metastases.

Study Population: Patients with advanced HCC who have:

* Confirmed extrahepatic metastases
* No prior PD-L1 or bevacizumab therapy
* Age 18-75 years
* Child-Pugh A or B7 liver function
* ECOG performance status 0-1

Treatment Regimen:

* PD-L1 antibody: 1200mg every 3 weeks
* Bevacizumab: 15mg/kg every 3 weeks
* HAIC with FOLFOX regimen: Up to 6 cycles
* Treatment continues until disease progression or up to 24 months

Primary Endpoint:

-Objective Response Rate (ORR)

Secondary Endpoints:

* Disease Control Rate (DCR)
* Duration of Response (DOR)
* Progression-free Survival (PFS)
* Overall Survival (OS)
* Safety assessments
* Quality of life measurements

Study Design Details:

* Single-arm study using Simon's two-stage design
* First stage: 27 patients
* Second stage: 9 additional patients if first stage shows efficacy
* Total planned enrollment: 36 patients
* Study duration: October 2024 - July 2027

This study aims to evaluate whether adding HAIC to PD-L1 inhibitor plus bevacizumab immunotherapy can improve outcomes for advanced HCC patients with extrahepatic spread, who currently have limited treatment options. The trial will assess both efficacy and safety of this combination approach.

ELIGIBILITY:
Inclusion Criteria:

Signed written informed consent Histologically/cytologically confirmed hepatocellular carcinoma (HCC) or clinically diagnosed according to HCC diagnostic criteria Radiologically confirmed extrahepatic metastases with unresectable disease as evaluated by investigators No prior treatment with PD-L1 antibody and/or bevacizumab Age ≥18 and ≤75 years ECOG Performance Status 0-1 Child-Pugh Class A or B7 Able to comply with study protocol requirements At least one measurable or evaluable lesion according to RECIST v1.1

Adequate organ and bone marrow function:

Absolute neutrophil count ≥1.5×10^9/L Platelet count ≥75×10^9/L Hemoglobin ≥9.0 g/dL Total bilirubin ≤2×ULN ALT and AST ≤5×ULN Serum creatinine ≤1.5×ULN or creatinine clearance ≥50mL/min Urine protein <2+ by dipstick APTT and INR ≤1.5×ULN Normal cardiac enzymes Normal thyroid function or on stable replacement therapy Life expectancy ≥12 weeks Effective contraception for participants of childbearing potential during treatment and for 6 months after last dose

Exclusion Criteria:

Severe complications from liver disease (severe bleeding from portal hypertension, infection, hepatic encephalopathy) Prior systemic anti-tumor therapy for HCC Other malignancy within 5 years (except adequately treated non-melanoma skin cancer or carcinoma in situ) Current participation in other interventional clinical trials Systemic treatment with Chinese herbal medicine or immunomodulators within 2 weeks before first dose Active autoimmune disease requiring systemic treatment within 2 years Systemic corticosteroid therapy within 7 days before first dose Prior allogeneic organ transplantation (except corneal) or stem cell transplantation Known allergy to monoclonal antibodies or HAIC components Inadequate recovery from prior treatment toxicities Known HIV infection Untreated active HBV infection (HBsAg positive with HBV-DNA above upper limit of normal) Active HCV infection Live vaccine administration within 30 days before first dose Pregnancy or breastfeeding

Serious or uncontrolled systemic diseases including:

Significant cardiac arrhythmias or conduction abnormalities Unstable angina or NYHA class ≥2 heart failure Arterial thrombotic events within 6 months Uncontrolled hypertension Active interstitial lung disease Active tuberculosis Active systemic infections Active diverticulitis or GI obstruction Uncontrolled diabetes Significant proteinuria Psychiatric disorders affecting compliance Any condition that could interfere with study participation or interpretation of results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by RECIST v1.1 | From first dose until disease progression or up to 24 months of treatment, with tumor assessments performed every 9 weeks for the first 48 weeks and every 12 weeks thereafter.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided